CLINICAL TRIAL: NCT06008002
Title: Evaluation of the Efficacy of M-TAPA and EXORA Block Application for Analgesia After Laparoscopic Cholecystectomy; Prospective, Single-blind, Observational Study
Brief Title: Evaluation of the Efficacy of Regional Anaesthesia for Analgesia After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-3/1
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Laparoscopic Cholecystectomy; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: prospective, single-blind, observational study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group M (Active Comparator): ultrasound guided Modified thoracoabdominal nerves block through perichondrial approach(M-TAPA) block
  Interventions: Procedure: M-TAPA block; Drug: Tramadol
- Group E (Active Comparator): Ultrasound guided External Oblique And Rectus Abdominis Plane (EXORA) Block
  Interventions: Procedure: EXORA block; Drug: Tramadol
- Group P (Active Comparator): Patient-controlled analgesia with tramadol
  Interventions: Drug: Tramadol

INTERVENTIONS:
Procedure: M-TAPA block — ultrasound guided Modified thoracoabdominal nerves block through perichondrial approach(M-TAPA) block (0.3 ml/kg , %0.25 bupivacaine) will be performed
  Arms: Group M
Procedure: EXORA block — Ultrasound guided External Oblique And Rectus Abdominis Plane (EXORA) Block block (0.3 ml/kg , %0.25 bupivacaine) will be performed
  Arms: Group E
Drug: Tramadol — 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; Patient-controlled analgesia settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.

SUMMARY:
Postoperative pain is important for patient comfort, wound healing and earlier mobilisation. Different procedures are used by clinicians for this purpose. Intravenous and regional anaesthesia techniques can be used for this purpose in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
In our study, the investigators aimed to investigate the effectiveness of different methods applied for post-operative pain in patients undergoing laparoscopic cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic cholecystectomy surgery
* Patients with ASA (American Society of Anaesthetists) scores I and III will be included.

Exclusion Criteria:

* Uncontrolled Arterial Hypertension
* Uncontrolled Diabetes Mellitus,
* Mental retardation ,
* Antidepressant use
* Metabolic disorders,
* Bleeding diathesis
* Patients with a body mass index above 30.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
NRS | Postoperative 24 hours
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
tramadol consumption | Postoperative 24 hours
side effect profile scores | Postoperative 24 hours
  1. Nausea and vomiting scale (nausea-vomiting scale (NVS):
  1. No nausea is present,
  2. Mild nausea is present.
  3. Severe nausea is present.
  4. Vomiting is present) In case of a NVS score of >3, an anti-emetic drug was administered.
additional analgesic use | Postoperative 24 hours
  additional analgesic use
pinprick test | Postoperative 24 hours
  The level of sensory block will be evaluated by pinprick test at 30 minutes following the block procedure and in postoperative patients.
  With the pinprick, the gently touches the skin with the pin or back end and asks the patient whether it feels sharp or blunt.
Ramsay Sedation Scale | Postoperative 24 hours
  Ramsay Sedation Scale (RSS) :
  1. Anxiety, agitation are present;
  2. Cooperated,awake;
  3. Sedated , response to commands;
  4. Sleepy, immediately awoken by auditory stimulus or glabella tap;
  5. Sleepy, deep response to auditory stimulus or glabella tap and
  6. Sleepy, no response to auditory stimulus or glabella tap )

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No